CLINICAL TRIAL: NCT07058025
Title: Mesenchymal Stromal Cells in Extreme Preterm Infants at Risk of Developing Bronchopulmonary Dysplasia - A Phase 2 Multi-Centre Double Blind Randomized Controlled Trial
Brief Title: Mesenchymal Stromal Cell Therapy to Prevent Bronchopulmonary Dysplasia in Extreme Preterm Infants
Acronym: HULC-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Stem Cell Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HULC-2
Record Dates: First submitted 2025-05-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Bronchopulmonary Dysplasia (BPD); ELGAN (22-28SA)
Keywords: Phase II clinical trial; Mesenchymal stromal cell; Cell therapy; Preterm infant; Bronchopulmonary Dysplasia; Extremely low gestational age neonates
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Intervention group:
  Participants allocated in the intervention group will receive multidose of UC-MSCs as follow:
  * Dose: each dose consists of 10x106 cells/kilograms of bodyweight.
  * Administration protocol: weekly IV dose of UC-MSCs for 3 weeks (total of 3 doses)
  * Route of administration: IV infusion on peripheral intravenous catheter. The UC-MSC solution will be infused using a syringe pump over 15 minutes, and after the UCMSC infusion, an additional volume of normal saline will be infused using a syringe pump over 15 minutes.
  Control group:
  Participants allocated in the control group will receive a sham procedure weekly for 3 weeks. A syringe of normal saline brought to bedside, but it will not be administered. The physician and bedside nurse will perform the sham procedure behind a screen (they will mimic IV catheter insertion and cell product injection)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parents of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group will receive multiple IV doses of UC-MSCs (Experimental): * Dose: each dose consists of 10 million cells/kilograms of bodyweight.
  * Administration protocol: weekly (7 days ± 1 day) IV dose of UC-MSCs for 3 weeks (Total of 3 doses)
  * Route of administration: IV infusion on peripheral intravenous catheter. The UC-MSC solution will be infused using a syringe pump over 15 minutes, and after the UCMSC infusion, an additional volume of normal saline will be infused over 15 minutes.
  Interventions: Biological: Human Allogenic Umbilical Cord Mesenchymal Stromal Cells
- Control group (Sham Comparator): Participants allocated in the control group will receive a sham procedure weekly for 3 weeks. A syringe of normal saline brought to bedside, but it will not be administered. The physician and bedside nurse will perform the sham procedure behind a screen (they will mimic IV catheter insertion and cell product injection)
  Interventions: Other: Sham procedure control

INTERVENTIONS:
Biological: Human Allogenic Umbilical Cord Mesenchymal Stromal Cells — IV administration of uc-MSC every 7 days ± 1 day for 3 weeks. Randomized double blinded
  Other Names: UC-MSC; Umbilical Cord Mesenchymal Stromal Cells; Mesenchymal Stromal Cells
  Arms: Intervention group will receive multiple IV doses of UC-MSCs
Other: Sham procedure control — Sham procedure (mimic IV catheter insertion adn cell product infusion behing a screen). Repeated weekly for 3 weeks
  Arms: Control group

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of mesenchymal stromal cell (MSC) therapy in extreme preterm infants to prevent bronchopulmonary dysplasia, the main respiratory complication of preterm birth.

Study participants will receive either multiple intravenous doses (total of 3 doses) of MSC derived from human donor umbilical cord tissue (intervention group) or no uc-MSC injection (control group) to confirm the safety of IV MSC in extreme preterm infants and evaluate the potential benefit of MSC therapy on their respiratory health as well as on other complications related to preterm birth.

DETAILED DESCRIPTION:
Include Background...

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) less than 28+0 weeks
* Post-natal age between 4 and 14 days of life
* Invasive ventilation with oxygen requirement:

  * On mechanical ventilation: intubated patient with any of the following ventilation modes: conventional, HFO or Jet ventilation:
  * With requirement of FiO2: FiO2 >= 30% and for at least 12 hours over 24 hours (i.e. flowsheets, FiO2 histogram)

Exclusion Criteria:

1. Congenital anomaly:

   * Genetic and chromosomal syndromes (e.g., Trisomy 13, Trisomy 18, Trisomy 21): either patient with high suspicion (antenatal findings, clinical features) or documented syndrome by genetic testing.
   * Major congenital anomalies including cardiac (i.e., congenital heart defects, NB. PDA is not considered an exclusion criterion), neurological (e.g., holoprosencephaly, anencephaly), gastrointestinal (e.g., gastroschisis, omphalocele), pulmonary (e.g., congenital diaphragmatic hernia) anomalies.
   * Inborn errors of metabolism.
2. Hemodynamic instability (shock):

   * Hemodynamic instability with impaired end-organ perfusion (metabolic acidosis with increased lactate and/or decreased urine output).
   * Requirements for fluid bolus, inotrope or vasopressor medication
3. Severe sepsis:

   * Signs of hemodynamic instability and requiring at least one fluid bolus.
   * And a positive blood or cerebrospinal fluid culture.
4. Pneumothorax: Pneumothorax with a chest tube in place
5. Severe pulmonary hemorrhage:

   * Active pulmonary hemorrhage (i.e., frank blood coming from the endotracheal tube.
   * And at least one of the following criteria: a)hemodynamic instability. b) blood product transfusion (packed red blood cells, platelets, fresh frozen plasma)
6. Extubation: If Extubation planned within the next 24 hours (post first uc-MSC administration/sham procedure).
7. Patient is not expected to survive:

   * Redirection of care.
   * Patient is moribund

Ages: 4 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2038-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of mechanical ventilation-free days accounting for mortality | 120 days
  The study primary outcome is the number of mechanical ventilation-free days accounting for mortality. Mechanical ventilation is defined by artificial ventilation using an endotracheal tube. For study purpose, this outcome will be measured at 120 days after randomization. To account for mortality, any death within 120 days post randomization will be counted as "0" mechanical ventilation-free day (worse outcome).

SECONDARY OUTCOMES:
Effects of uc-MSCs on the date of extubation for participants. | From date of randomization until the date of discharge home or date of death from any cause, whichever came first, assessed up to 12 months
  This respiratory outcome will be measured to determine if uc-MSCs have an effect on the date of extubation for participants
Effects of uc-MSCs on the rate of survival without moderate or severe BPD at 36 weeks corrected age. | BPD severity will be assessed for each participant at 36 weeks of corrected age
  This will assess if uc-MSCs impact survival with moderate or severe Bronchopulmonary dysplasia.
Effects of uc-MSCs on the Number of Participants receiving open-label dexamethasone for severe chronic lung disease | From date of randomization until the date of discharge home or date of death from any cause, whichever came first, assessed up to 12 months
  This will help us determine if the intervention reduces use of dexamethasone for the treatment of severe chronic lung disease.
Effects of uc-MSCs on the duration of respiratory support. | From date of randomization until the date of discharge home or date of death from any cause, whichever came first, assessed up to 12 months
  Since ventilation damages underdeveloped lungs, determining the duration of ventilation is important to monitor as an outcome of uc-MSCs.
  We will collect the total number of days on mechanical ventilation, non-invasive ventilation, and oxygen therapy during the NICU hospitalization for each participant
Effects of uc-MSCs on the levels of respiratory support at 36 weeks CA, 40 weeks CA and at hospital discharge. | From date of randomization until the date of discharge home or date of death from any cause, whichever came first, assessed up to 12 months
  The different levels of intensity of ventilation will help us determine if uc-MSCs reduce ventilation days.
  The respiratory support being used are the following (Room air being the least intensive and best for participant health outcome.):
  mechanical ventilation vs. Continuous Positive Airway pressure/High Flow Nasal Canula, vs. Low Flow Nasal Canula vs. room air
Effects of uc-MSCs on the occurrence of pulmonary hypertension related to severe BPD | From date of randomization until the date of discharge home or date of death from any cause, whichever came first, assessed up to 12 months
  This will help us determine the therapeutic properties of UC-MSCs in reducing the occurrence of pulmonary hypertension related to severe BPD.
  Participants will be screened by echocardiography for pulmonary hypertension at 36 weeks of corrected age. Medication for chronic pulmonary hypertension will be collected.
Neurodevelopment and health outcomes at 24 months corrected age (Bayleys) | Assessment will be scheduled at 24 months corrected age.
  The neurodevelopmental assessment will be scheduled at 24 months CA with a window of +/- 6 months (i.e., between 18 to 30 months CA). Participants will be evaluated in the Neonatal Follow-Up clinic for high-risk infants. An assessment of general health and growth will be performed, and the most recent audiology and ophthalmology results will be recorded. The Bayley Scales of Infant Develpment-4th edition will be performed by a qualified professional to further evaluate the neurodevelopment of the participant.
Evaluation of safety of IV administration of UC-MSCs: Dose Limiting toxicity | 24-hours post uc-MSC injection
  Dose-limiting toxicity, defined as one of the following events, occurring within 24-hour post UC-MSC injection:
  * Death
  * Anaphylaxis
  * Increase need for respiratory support define by increase FiO2 >30% from baseline and/or increase in mean airway pressure > 5 cmH2O from baseline
  * Medications to support hemodynamic status (including management of cardiac arrest) including fluid boluses, inotropes, or vasopressors
  * Any SAE not expected in this patient population for which there is no alternative explanation but the IV administration of UC-MSCs and occurring within 1 week after UC-MSCs injection.
Evaluation of safety of IV administration of UC-MSCs: potential adverse event | within 1 week post uc-MSC injection
  Any Serious Adverse Event (SAE) not expected in this patient population for which there is no alternative explanation but the IV administration of UC-MSCs and occurring within 1 week after UC-MSCs injection.
Long-term participant safety follow-up | From enrollment until participant is 10 years of age.
  We plan to have annual parental interviews via telephone until the participant is 10 years old. This is to assess the respiratory status and any new diagnoses of study participants.
Complications of prematurity (assessed at time of hospital discharge) | From date of randomization until the date of discharge home or date of death from any cause, whichever came first, assessed up to 12 months
  The complications of prematurity assessed are the following:
  * BPD.
  * Patent Ductus Arteriosus requiring medical, surgical or device closure.
  * Intra-ventricular hemorrhage ≥ grade 3 according to Papille's classification.
  * Periventricular leukomalacia.
  * Necrotizing enterocolitis ≥ stage 2 according to Bell's classification.
  * Retinopathy of prematurity requiring treatment
  * Late-onset sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Thébaud, MD, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (8):
- Canada (8):
  - Royal Alexandra Hospital/Stollery Children's Hospital, Edmonton, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Ctr, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - McGill Montreal Children's Hospital, Montreal, Quebec
  - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No